CLINICAL TRIAL: NCT07405255
Title: Clinical Study on the Efficacy and Safety of Zanubrutinib Combined With Chemotherapy for Continuous Maintenance Treatment of Newly Diagnosed Central Nervous System Lymphoma
Brief Title: Zillion: Zanubrutinib Combined With Chemotherapy for Newly Diagnosed CNS Lymphoma
Acronym: Zillion
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, prof, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zillion
Record Dates: First submitted 2025-08-08; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Central Nervous System Lymphoma
MeSH Terms: interventions — zanubrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm: Zanubrutinib + Rituximab + MTX ± Selinexor (Experimental): This single treatment arm includes an induction phase of six 21-day cycles where participants receive:
  Zanubrutinib 160 mg orally twice daily, Rituximab 375 mg/m² intravenously on Day 0, MTX 3.5 mg/m² intravenously on Days 1.
  Before starting the second cycle, TP53 mutation status will be assessed. Participants positive for TP53 mutation will have Selinexor 60 mg orally added on Days 1 and 3 weekly.
  Following induction, a maintenance phase consists of Zanubrutinib 160 mg orally twice daily for up to 2 years or until disease progression or unacceptable toxicity.
  This study uses a biomarker-driven approach within a single-arm design without randomization or comparator arms.
  Interventions: Drug: Zanubrutinib + Rituximab + MTX ± Selinexor

INTERVENTIONS:
Drug: Zanubrutinib + Rituximab + MTX ± Selinexor — This is a single-arm interventional study. Participants will undergo an induction phase consisting of six 21-day cycles. During induction, all participants receive:
  Zanubrutinib 160 mg orally twice daily, Rituximab 375 mg/m² intravenous on Day 0, MTX 3.5 mg/m² intravenous on Days 1.
  Before the second treatment cycle, participants will be tested for TP53 mutation status. Participants who test positive for the TP53 mutation will receive Selinexor 40 mg orally on Days 1 weekly added to their treatment regimen.
  Following induction, participants enter a maintenance phase with:
  Zanubrutinib 160 mg orally twice daily, continued for up to 2 years or until disease progression or unacceptable toxicity.
  This design allows biomarker-driven treatment modification within a single treatment arm without randomization or separate comparator groups.

SUMMARY:
Subjects who met the inclusion/exclusion criteria were included in the experimental group after signing the informed consent form. One course of Z(R)-MTX(TMZ) treatment was given. After the results of the second-generation sequencing were reported, selinisol was added to the original treatment plan for those with TP53 mutations, and the original treatment plan was continued for those without TP53 mutations. Each course of treatment lasts for three weeks. A mid-term assessment is conducted after three courses of treatment, and a final assessment is carried out after six courses of treatment. After the mid-term or final assessment:

If the PR is not achieved or the disease progresses at any time, the subjects are withdrawn from the group and receive salvage treatment.

If the subjects achieve CR or PR, they enter maintenance treatment and continue with zanubrutinib for 2 years. For young patients (< 65 years old), they can choose whether to receive ASCT as consolidation treatment according to their personal will, and then follow up and observe until 3 years have passed.

SD/PD patients receive subsequent treatment after being judged by the researchers

ELIGIBILITY:
Inclusion Criteria:

* Have a full understanding of this study and voluntarily sign the informed consent form.
* Untreated patients with primary central nervous system lymphoma (PCNSL) confirmed by pathology (immunotyping) according to the 2016 WHO classification of lymphoid neoplasms.
* Diffuse large B-cell lymphoma (DLBCL) originating from the central nervous system (CNS) without involvement of other organs, confirmed by PET-CT or contrast-enhanced CT.
* Expected survival greater than 3 months.
* Laboratory test results meeting all of the following:
* Creatinine clearance rate ≥ 50 mL/min (calculated by the Cockcroft-Gault formula).
* International normalized ratio (INR) ≤ 1.5 × ULN or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN. Patients on warfarin may have INR 2-3.
* Left ventricular ejection fraction (LVEF) ≥ 50%.
* Glomerular filtration rate (GFR) ≥ 60 mL/min.
* Male or female patients of childbearing potential must agree to use effective contraception (e.g., double-barrier methods, condoms, oral or injectable contraceptives, intrauterine device) during the study and for 30 days after the last dose.
* Postmenopausal women (> 45 years old and amenorrheic > 1 year) or surgically sterilized women are exempt from this requirement.

Exclusion Criteria:

* Contraindication to any drug included in the treatment regimen.
* History of clinically significant liver disease, including viral or other hepatitis or cirrhosis.
* Hepatitis B: Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with HBV-DNA above ULN.
* Active hepatitis C: Positive HCV antibody with detectable HCV-RNA.
* Human Immunodeficiency Virus (HIV) infection.
* Congestive heart failure (New York Heart Association Class > II) or history within 6 months of acute myocardial infarction, unstable angina, stroke, or transient ischemic attack.
* Hereditary long QT syndrome or QTc > 480 ms (QTc calculated using Fridericia's formula, QTcF = QT / RR^0.33).
* Other malignancies within 5 years, except: completely cured cervical carcinoma in situ, basal cell carcinoma of the skin, breast carcinoma in situ, or another primary cancer that has been cured and not recurred within 5 years.
* Pregnant or lactating women, or women planning pregnancy during the study period.
* History of significant neurological or psychiatric disorders, including substance or psychotropic-drug abuse.
* Clinically significant active infection.
* Inability to take or swallow oral medication, or conditions affecting drug absorption (e.g., chronic diarrhea, intestinal obstruction).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete Remission Rate (CRR) | At the end of Cycle 6 and at 4 weeks after completion of Cycle 6 (each cycle is 21 days).
  Complete Remission Rate (CRR) is defined as the proportion of participants achieving complete remission based on predefined hematologic and/or imaging criteria at the end of treatment Cycle 6.

SECONDARY OUTCOMES:
Overall Survival (OS) | From initiation of study treatment to death from any cause or last follow-up, whichever occurs first, up to 2 years.
  Overall Survival (OS) is defined as the time from initiation of study treatment to death from any cause. Participants who are alive at the time of analysis will be censored at the date they were last known to be alive. OS will be summarized using the Kaplan-Meier method.

OTHER OUTCOMES:
Number of participants with treatment-related Adverse Events (AEs) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | From initiation of study treatment through the end of treatment (up to 6 cycles; each cycle is 21 days).
  Safety will be evaluated by monitoring and recording the number, type, and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The number of participants experiencing treatment-related AEs will be summarized by frequency and grade.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China